CLINICAL TRIAL: NCT06091228
Title: The Additional Effect of Including Tongue Scraping to the Oral Hygiene Instructions on Halitosis Parameters in Periodontitis Patients Undergoing Standard Initial Periodontal Therapy
Brief Title: The Additional Effect of Tongue Scraping on Halitosis Parameters in Initial Periodontal Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Ana CASTRO SARDA, Dr, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S67590
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Periodontitis; Halitosis; Tongue Condition
Keywords: periodontitis; halitosis; oral malodor; tongue coating; tongue cleaning; non-surgical treatment
MeSH Terms: conditions — Periodontitis; Halitosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control- No tongue scraping full length of study (No Intervention): Oral hygiene instructions before and after non-surgical treatment without inclusion of tongue scraper
- Test 1 - tongue scraping full length of study (Experimental): Oral hygiene instructions before and after non-surgical treatment with inclusion of tongue scraper
  Interventions: Other: tongue scraper
- Test 2 - tongue scraping only after non-surgical therapy (Experimental): Oral hygiene instructions before and after non-surgical treatment with inclusion of tongue scraper only after treatment
  Interventions: Other: tongue scraper

INTERVENTIONS:
Other: tongue scraper — tongue cleaning with gentle strokes twice a day covering the whole surface of the tongue
  Arms: Test 1 - tongue scraping full length of study; Test 2 - tongue scraping only after non-surgical therapy

SUMMARY:
Periodontitis can lead to tooth loss which may impair chewing ability and aesthetics. In addition, periodontitis can give rise to halitosis.

Standard initial periodontal treatment consists of supra and subgingival biofilm reduction and removal of calculus. Recently, the European Federation of Periodontology introduced clinical practice guidelines for the treatment of periodontitis. The use of a tongue scraper is not mentioned as element in the standard initial treatment of periodontitis.

We have planned a clinical study in order to provide information about the effect of standard initial periodontal therapy and the additional effect of the use of a tongue scraper as part of the oral hygiene instructions on halitosis parameters in periodontitis patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures 2. Males or females American Society of Anesthesiologist classification I of II, 3. 18 years of age or older, 4. In good general health as documented by self-assessment 5. Suffer from generalised periodontitis (according to 2018 classification) 4 6. Suffer from halitosis with suspected intra-oral cause: organoleptic score of 2 or higher by an experienced oral malodour judge 7. At least one volatile sulphur compounds measurement above the following thresholds:

  1. Portable sulphur detector > 107 ppb 26
  2. Oral Chroma™: hydrogen sulfide (H₂S) > 112ppb
  3. Oral Chroma™: methyl mercaptan (CH3SH) >28ppb (as recommended by manufacturer).

Exclusion Criteria:

* 1. Participant has a history of chemotherapy or radiotherapy in head and neck area 2. Any disorder, which in the Investigator's opinion might jeopardise the participant's safety or compliance with the protocol 3. Any prior or concomitant treatment(s) that might jeopardise the participant's safety or that would compromise the integrity of the Trial 4. Female who is pregnant, breast-feeding or has the intention of becoming pregnant in the following 6 months 5. Participation in another interventional Trial with an investigational medicinal product (IMP) or device 6. Recent intake of antibiotics (3 months prior to the first consultation) 7. Antibiotics indicated as part of the periodontal treatment 8. Use of antibiotics during the course of the study 9. Suffer from halitosis with suspected extra-oral cause 10. Suffer from a systemic disease that could cause extra-oral halitosis (e.g. diabetes mellitus, liver or kidney failure, trimethylaminuria) 11. Participant has a history of rheumatic fever, neurological deficiencies, or use of medication which may affect periodontal tissue, (phenytoin, cyclosporin, nifedipine, chronic use of non-steroidal anti-inflammatory drugs) 12. Presence of active caries lesions 13. Unwillingness to return for the follow-up examination 14. Wear partial prosthetic dentures removables 15. Participant has less than 20 teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Improving of halitosis parameters (organoleptic scores) | 18 weeks
  reduction in scores

SECONDARY OUTCOMES:
improving of volatile sulphur compounds | 18 weeks
  reduction in ppb
improving of periodontal parameters | 18 weeks
  reduction in pocket depth
improving of oral hygiene parameters. | 18 weeks
  reduction in full mouth bleeding score and full mouth plaque score

CONTACTS AND LOCATIONS:
Overall Officials: Ana Castro, Principal Investigator — Universitaire Ziekenhuizen KU Leuven

IPD SHARING:
Plan to Share IPD: No